CLINICAL TRIAL: NCT02017600
Title: A Phase II Trial of Induction Chemotherapy With ND-420, Cisplatin and Fluorouracil Followed by Surgery in the Treatment of Patients With Localized Squamous Cell Carcinoma of the Esophagus
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Nang Kuang Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NKCND420/201112
Record Dates: First submitted 2013-12-09; First posted 2013-12-23 (Estimated); Last update posted 2020-05-20 (Actual); Status verified 2020-05

CONDITIONS: Localized Squamous Cell Carcinoma of the Esophagus
MeSH Terms: interventions — Surgical Procedures, Operative; Cisplatin; Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Induction Chemotherapy DCF followed by Surgery (Experimental): All eligible patients will receive ND-420, Cisplatin and fluorouracil every 3 weeks for 2 cycles. After induction chemotherapy, patients will be planned to receive Surgery.
  Interventions: Drug: ND-420; Procedure: Surgery; Drug: Cisplatin; Drug: fluorouracil

INTERVENTIONS:
Drug: ND-420 — ND-420 50 mg/m2 on day1
  Other Names: ND-420(Nangkuang)
Procedure: Surgery — After induction chemotherapy, participants will be receive right or left thoracotomy for curative resection by total or subtotal thoracic esophagectomy.
Drug: Cisplatin — cisplatin 70 mg/m2 on day1
Drug: fluorouracil — fluorouracil 700 mg/m2 daily, day1 to day4
  Other Names: 5-FU

SUMMARY:
Investigator will assign 53 patients who had been histologically proven localized squamous cell carcinoma of esophagus to receive the induction chemotherapy regimen of ND-420 50 mg/m2 on day 1, cisplatin 70 mg/m2 on day1, plus fluorouracil 700 mg/m2 daily, day1 to day4, every 3 weeks for 2 cycles and then followed by surgical resection. The successful rate of complete treatment per protocol and complete resection will be the primary variant to evaluate in our study.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have been histologically proven esophageal carcinoma (squamous cell carcinoma).
* The tumor had to be locally advanced (stage T2-3/N0, T1-3/N+, if technically resectable with curative intent).
* Patients must be 20 years of age.
* Patients must have an ECOG performance status score 2.
* Patients must have a life expectancy of at least 12 weeks.
* Patients must be accessible for treatment and follow-up at least for one year.
* Patients must sign the informed consent form.
* Patient must have:Hemoglobin level 9 g/dl; Neutrophil count 1,500/mm3; Platelets count 100,000/mm3; Serum bilirubin level 1.0 ULN; Serum transaminase (GOT, GPT) levels 2.0 ULN; Serum Alkaline phosphatase levels 2.0 ULN; Serum creatinine level 1.5 mg/dl or Creatinine clearance rate(CrCl)60 ml/min for the institution (calculated by the Cockcroft- Gault equation).

Exclusion Criteria:

* Patient who are receiving or had received concurrent radiotherapy, chemotherapy or other anticancer treatment for esophageal carcinoma.
* Patients with known history of severe hypersensitivity reactions to any medicine or to drugs formulated with polysorbate 80.
* Major surgery within two weeks prior to entering the study, excluding port-A insertion or feeding jejunostomy surgery.
* Patients with CNS metastasis, including clinical suspicion.
* Patients with clinically detectable peripheral neuropathy 2 on the CTC criteria.
* Mental statuses of patients are not fit for clinical trial.
* Fertile men and women unless using a reliable and appropriate contraceptive method.
* Patients with pregnancy or lactating, women considering pregnancy, possible pregnancy that without using effective contraception.
* Patients who have serious concomitant illness that might be aggravated by chemotherapy, as below included:Active cardiac disease (e.g. congestive heart failure, angina, arrhythmia, acute myocardial disease or other types of heart disease requiring treatment) within 6 months period preceding entry into the study; Uncontrolled infection (e.g. active infection that uncontrolled for 2 weeks under antibiotic therapy); Retention of body fluid (e.g. pleural effusion, ascites, pericardial effusion, and edema needing treatment); History of other than esophageal cancer, except curatively treated non-melanoma skin cancer or in situ carcinoma of the esophagus; and other conditions which will be judged by physician's discretion.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2013-08; Primary Completion 2014-12-02 (Actual); Study Completion 2015-04-04 (Actual)

PRIMARY OUTCOMES:
the R0 resection rate of participants | up to three months

SECONDARY OUTCOMES:
the response rate (RECIST) of participants | up to three months
Number of participants with adverse events as a measure of safety and tolerability | up to one year
the population pharmacokinetic parameters (Cmax, AUC... )of ND-420 in the participants | 0, 30min, 1hr of ND-420 infusion. selected randomly form one of 3hr, 7hr, 11hr and 23hr after the end of ND-420 infusion.
the correlation between clinical outcomes and the potential predictive genomic biomarkers(B-tubulin mutation, p53-Arg 72Pro, Bcl2-C938A, MDR1-C3435T polymorphism, TNFRSF1B-1466, GSTP1-l105V, CYP1B1, TS-5'UTR) for tumor response | up to one year
1-year survival rate of participants | up to one year
pathologic complete response rate of participants | up to one year
1-year progression free survival rate of participants | up to one year
1-year overall survival rate of participants | up to one year

CONTACTS AND LOCATIONS:
Overall Officials: Ming-Huang Chen, M.D., Principal Investigator — Taipei Veterans General Hospital, Taiwan
Locations (1):
- Taipei Veterans General Hospital, Taipei, Taiwan